CLINICAL TRIAL: NCT01372969
Title: Multicenter Phase I/IIa Study to Assess the Safety and Efficacy of Expanded Allogenic Adipose-derived Stem Cells (eASCs) (Cx601), for Treatment of Complex Perianal Fistulas in Perianal Crohn's Disease.
Brief Title: Study to Assess the Safety and Efficacy of Expanded Allogenic Adipose-derived Stem Cells (eASCs) (Cx601), for Treatment of Complex Perianal Fistulas in Perianal Crohn's Disease.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cx601-0101
Record Dates: First submitted 2010-08-30; First posted 2011-06-14 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease; Anal Fistula
MeSH Terms: conditions — Crohn Disease; Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cx601 (Experimental)
  Interventions: Drug: Cx601

INTERVENTIONS:
Drug: Cx601 — Suspension of adult expanded allogenic adipose-derived stem cells (eASCs) at a doses of 20 million cells and 40 million cells.

SUMMARY:
The purpose of this study is to asses the safety and efficacy of adipose-derived adult stem cells from healthy donnors for treatment of complex perianal fistulas in Crohn's disease.

DETAILED DESCRIPTION:
Crohn´s disease (CD) is a severe disorder with significant morbidity and major impact on life. CD can affect any part of the digestive system and symptoms of this chronic illness include abdominal pain, bloating, nausea, vomiting and diarrhea. CD also causes bowel wall ulcers, strictures (narrowing of a hollow structure due to scar tissue and swelling), and fistulas (abnormal passages from the intestines to another organ or the skin).

There is an unmet need for effective medical therapy in CD patients with perianal fistulas, not responding to the conventional strategies, including biological therapies. The current study is designed to assess the safety and efficacy of adipose tissue derived mesenchymal stem cells from healthy donors for the treatment of perianal fistulas in patients presenting CD.

Primary objective: To assess the safety (incidence of treatment emergent adverse-events) of eASCs.

Study design: Multicenter, pilot study, assessing safety and with evaluation of the efficacy by two Gastroenterologists/Surgeons and an independent external radiologist. Subjects will receive a cell suspension of allogenic adipose-derived stem cells, eASCs (20 million cells) in the fistula.

In case of incomplete fistula closure of the treated fistula at week 12, subjects will receive a second dose of eASCs (40 million cells). Subjects will be followed until week 24, following the initial administration of cells.

Subjects may be treated with standard care during the entire study period, according to the investigators discretion, excluding infliximab or any other anti-TNF, tacrolimus or cyclosporine.

. Study population: In total 24 patients, men and women of at least 18 years of age, with perianal CD will be recruited. Patients with a minimum of one and a maximum of three fistula tracts.

Description of treatments: .

Subjects will receive:

Investigational product: CX-601 Suspension of adult expanded allogenic adipose-derived stem cells (eASCs) at a doses of 20 million cells and 40 million cells.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Subjects with Crohn's disease diagnosed at least 12 months earlier in accordance with accepted clinical, endoscopic, anatomopathological and/or radiologic criteria.
* Presence of complex perianal fistula with 3 or fewer fistulous tracts assessed by MRI,
* Subjects with persistent and active complex perianal fistula and non active luminal CD defined by a CDAI ≤ 200.
* Subjects of either sex aged over 18 years. Good general state of health according to the findings of the clinical history and the physical examination.

Exclusion Criteria:

* Presence of severe proctitis (prominent friability, spontaneous bleeding, multiple erosions, deep ulcers) or dominant active luminal disease requiring immediate therapy, assessed by rectosigmoidoscopy
* Subjects with a CDAI ≥ 221.
* Subjects with an abscess (unless a complete toilet of the area with drainage of the collections and the absence of abscess and other collections is confirmed prior to treatment start).
* The presence of setons unless removed prior to treatment start.
* Presence of >3 fistulous tracts and/or external openings.
* Subjects with rectal and/or anal stenosis evaluated by rectoscopy or EUA.
* Subjects who have received infliximab or any other anti-TNF agent in the 8 weeks before the cell treatment administration.
* Subjects who have received tracrolimus or ciclosporine in the 4 weeks before the cell treatment administration.
* Subjects with rectovaginal fistula, anal fistula(s), and/or non-perianal enterocutaneous fistula.
* Subjects with a history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion.
* Subjects with malignant tumor, except for basal cell or cutaneous squamous cell carcinoma, or Subjects with a prior history of malignant tumors, unless the neoplastic disease has been in remission for the previous 5 years.
* Subjects with cardiopulmonary disease which, in the opinion of the investigator, is unstable or sufficiently serious to exclude the patient from the study.
* Subjects with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from the study.
* Subjects with congenital or acquired immunodeficiencies.
* Subjects with abnormal laboratory test findings that contraindicate their inclusion in the study.
* Subjects allergic to anesthetics or MRI contrast.
* MRI is unfeasible, (e.g. due to the presence of pacemakers, hip replacements or severe claustrophobia)
* Subjects in need of surgery in the perianal region for reasons other than fistulas at the time of inclusion in the study, or a need for such surgery is foreseen in this region in the 26 weeks after treatment administration.
* Subjects who have suffered major surgery or severe trauma in the prior 6 months.
* Pregnant or breastfeeding women. (Both men and women should use appropriate birth control methods defined by the investigator).
* Subjects currently receiving, or having received within 1 month prior to enrolment into this clinical trial, any investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse-events | 24 weeks

SECONDARY OUTCOMES:
The reduction in the number of draining fistulas | weeks 10,12, 22 and 24
The increase in the number of closed fistulas. | weeks 12 and 24
Percentage of subjects in whom, the external openings of treated perianal fistula have closed. | week 12
Percentage of subjects with MRI fistula healing (absence of collections >2cm) | weeks 12 and 24
Percentage of subjects presenting luminal relapse | weeks 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Damián García Olmo, MD, Principal Investigator — Hospital La Paz
Locations (6):
- Spain (6):
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital San Juan de Dios del Aljarafe, Bormujos, Sevilla
  - Hospital Juan Ramón Jimenez, Huelva
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Virgen de la Macarena, Seville